CLINICAL TRIAL: NCT01467063
Title: Dietary Amino Acids and Insulin Sensitivity in Children With Type 1 Diabetes
Brief Title: Glutamine and Insulin Sensitivity in Type I Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Dominique Darmaun, Prinicipal Investigator, Nemours Children's Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRC# 11-29
Record Dates: First submitted 2011-11-02; First posted 2011-11-08 (Estimated); Results first posted 2021-01-29 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Type I Diabetes Mellitus
Keywords: Type I Diabetes; Insulin Resistance; Glutamine; Amino Acids; Glucagon like peptide 1; Glutathione; Citrulline; Arginine; Nitric Oxide
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glutamine (Active Comparator)
  Interventions: Dietary Supplement: Glutamine
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Glutamine — Participants will keep a diary of food intake and activity as well as wear an accelerometer (to measure overall movement) for 2-3 days prior to the admission. Subject will come to the Clinical Research Center for approximately 24 hours. They will receive a drink containing Glutamine (0.25 g/kg/dose). Afterwards they will have an afternoon exercise session consisting of 15-min bouts of exercise, interspersed with 5-min rest periods in between for a total of 75min. Blood glucose will be checked during rest intervals. They will be served a controlled dinner. Before bedtime another dose of the same drink will be given. Overnight blood glucose will be monitored closely. In the morning, another dose of the same drink will be given. Subjects will have two isotope infusions (non-radioactive) running concomitantly and a hyperinsulinemic-euglycemic clamp will be performed. Afterwards lunch will be served and subject discharged home.
  Arms: Glutamine
Dietary Supplement: Placebo — Participants will keep a diary of food intake and activity as well as wear an accelerometer (to measure overall movement) for 2-3 days prior to the admission. Subject will come to the Clinical Research Center for approximately 24 hours. They will receive a PLACEBO drink. Afterwards they will have an afternoon exercise session consisting of 15-min bouts of exercise, interspersed with 5-min rest periods in between for a total of 75min. Blood glucose will be checked during rest intervals. They will be served a controlled dinner. Before bedtime another dose of the same drink will be given. Overnight blood glucose will be monitored closely. In the morning, another dose of the same drink will be given. Subjects will have two isotope infusions (non-radioactive) running concomitantly and a hyperinsulinemic-euglycemic clamp will be performed. Afterwards lunch will be served and subject discharged home.
  Arms: Placebo

SUMMARY:
Insulin is crucial to help the body metabolize ('burn') sugar (glucose). Even though juvenile (type 1) diabetes (T1D) is primarily due to the lack of insulin, patients with T1D tend to become less sensitive to insulin, particularly during adolescence.

The overall objective of this project is to gain further insight into the possible benefits of supplementation with glutamine (GLN), a natural dietary amino acid, enhancing insulin sensitivity in adolescents with T1D. To elucidate the impact of glutamine, the investigators will use a method called the 'euglycemic, hyperinsulinemic clamp': it consists of giving an IV drip of insulin, while the drop in blood sugar is prevented by giving variable, precisely measured amounts of glucose by vein: the amount of glucose required to prevent a drop in blood sugar reflects the body's sensitivity to insulin. The investigators will also give an IV drip of glucose and arginine (a building block of protein) 'tagged' with non-radioactive isotopes to better understand how glutamine may work. This procedure will be performed in 2 groups of 10 adolescents in the morning either after a strenuous exercise performed the previous afternoon (group 1; n=10), or after a sedentary day (group 2; n=10). Each subject will be studied twice, once after taking oral GLN, once after placebo, in separate clinical research center (CRC) admissions a few weeks apart, in random order.

Should the investigators hypothesis prove to be true, it would warrant long term studies to determine whether sustained dietary GLN supplementation can decrease insulin requirements and ultimately improve diabetes control in teenagers with T1DM, If successful, this approach could potentially have a significant positive impact in terms of adolescent health.

ELIGIBILITY:
Inclusion Criteria:

* Type I diabetes diagnosed for > 12 months.
* Minimal weight of 40 kg
* Tanner stage IV or beyond
* All insulin programs, including intermediate/short acting insulins, Lantus/Detemir and short acting insulin or insulin pump therapy.
* HbA1C between 7.5 and 10%
* BMI between 10th to 85th percentile
* Patients on stable thyroid replacement therapy will be allowed to participate.

Exclusion Criteria:

* Celiac disease (any patient with history of positive serology or consuming a gluten-free diet)
* Cystic Fibrosis
* Chronic steroid therapy
* Chronic medications that may interfere with glucose metabolism or liver function
* History of mental retardation
* Presence of diabetic complications
* Positive pregnancy test
* Presence of significant anemia (Hb<11 g/dL)
* Presence of intercurrent infection

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Darmaun, MD, PhD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

REFERENCES:
- [Background] Mauras N, Xing D, Fox LA, Englert K, Darmaun D. Effects of glutamine on glycemic control during and after exercise in adolescents with type 1 diabetes: a pilot study. Diabetes Care. 2010 Sep;33(9):1951-3. doi: 10.2337/dc10-0275. Epub 2010 Jun 28. PMID 20585005
- [Result] Torres-Santiago L, Mauras N, Hossain J, Weltman AL, Darmaun D. Does oral glutamine improve insulin sensitivity in adolescents with type 1 diabetes? Nutrition. 2017 Feb;34:1-6. doi: 10.1016/j.nut.2016.09.003. Epub 2016 Sep 20. PMID 28063503

RESULTS

PARTICIPANT FLOW:
Groups:
- Glutamine, Then Placebo; Placebo, Then Glutamine: Thirteen subjects were recruited, 12 of 13 completed the study; 2 did not receive isotope infusions but underwent all other procedures and were included in all analyses.
Period: Overall Study
Arm/Group | Glutamine, Then Placebo | Placebo, Then Glutamine
Started | 6 | 7
Completed | 5 | 7
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 16 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Insulin sensitivity as measured by hyperinsulinemic-euglycemic clamp. Insulin sensitivity was calculated by dividing the average glucose infusion rate (mL glucose infusion/kg body weight/min) by the average insulin concentration (uU/mL).
Time Frame: During the Hyperinsulinemic-Euglycemic Clamp, an average of 3 hours
Population: Thirteen subjects were recruited, 12 of 13 completed the study; 2 did not receive isotope infusions but underwent all other procedures and were included in all analyses.
Measure: Least Squares Mean (Standard Error); unit: mL/kg/min per uU/mL
Arm/Group | Glutamine | Placebo
Number analyzed (Participants) | 12 | 12
mL/kg/min per uU/mL | 0.1 (0.02) | 0.07 (0.02)

2. Secondary Outcome: Glucagon-like Peptide 1 (GLP-1)
Time Frame: Post-Infusion
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Glutamine | Placebo
Number analyzed (Participants) | 12 | 12
pmol/L | 2.3 (0.3) | 1.8 (0.1)

ADVERSE EVENTS:
Groups:
- Glutamine; Placebo: Thirteen subjects were recruited, 12 of 13 completed the study; 2 did not receive isotope infusions but underwent all other procedures and were included in all analyses.
Arm/Group | Glutamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No